CLINICAL TRIAL: NCT02826395
Title: Carbon-11 Sodium Acetate PET/CT Imaging of Prostate Cancer
Brief Title: C11 Sodium Acetate PET/CT Imaging of PCa
Status: No longer available | Type: Expanded Access
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ACETATE16-000260EA; 16-000260 (Other: UCLA/Jonsson Comprehensieve Cancer Center)
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; diagnostic; imaging; PET/CT; Acetate carbon-11
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — carbon-11 acetate

INTERVENTIONS:
Drug: Carbon-11 Sodium Acetate — PET/CT Scans will be performed with or without oral and IV contrast. All investigational scans will be read by at least one board-certified nuclear medicine physician with established expertise in PET/CT of at least 5 years' experience. Fifteen minutes after injection of 11C-Sodium Acetate, we will acquire a scan Emission images will be acquired for 3-5min/bed position. Intravenous and oral contrast will be given for the CT portion of the study.
  Other Names: C11 Sodium Acetate, C11 Acetate

SUMMARY:
The investigators propose to conduct Carbon-11 Sodium Acetate PET/CT studies. The purpose of our study is to evaluate the impact of Carbon-11 Sodium Acetate PET/CT studies on patient management in patients with prostate cancer.

DETAILED DESCRIPTION:
This is an expanded access study under an IND with a total of 300 participants with prostate cancer. Eligible participants will undergo baseline assessments at enrollment. Study participants will receive 11C-Sodium Acetate and will undergo a PET/CT imaging study. All patients referred by Oncologists and Urologists will be screened by a UCLA Nuclear Medicine physician and then accepted for scanning if clinically appropriate. The following steps will take place.

1. Informed consent will be obtained.
2. Vital signs (heart rate, blood pressure, respiratory rate, pulse oxymetry) will be recorded.
3. Participant will be injected with 20 - 40mCi of 11C-Sodium Acetate intravenously (i.v.).
4. PET/CT Scans will be performed with or without oral and IV contrast. All investigational scans will be read by at least one board-certified nuclear medicine physician with established expertise in PET/CT of at least 5 years' experience. Fifteen minutes after injection of 11C-Sodium Acetate, the investigators will acquire a scan. Emission images will be acquired for 3-5min/bed position. Intravenous and oral contrast will be given for the CT portion of the study.
5. Vital signs (heart rate, blood pressure, respiratory rate, pulse oxymetry) will be recorded following the completion of the scan.
6. Within 24-48 hours of PET/CT imaging, a follow-up telephone call or email will be conducted to discuss any side effects or reactions to the investigational agent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed prostate cancer
* Able to remain still for duration of each imaging procedure (about 30 minutes)

Exclusion Criteria:

* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.

Sex: Male
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- 200 Medical Plaza, B114, Los Angeles, California, United States

REFERENCES:
- [Background] Czernin J, Benz MR, Allen-Auerbach MS. PET Imaging of Prostate Cancer Using C-Acetate. PET Clin. 2009 Apr;4(2):163-72. doi: 10.1016/j.cpet.2009.05.001. No abstract available. PMID 21984877
- See also: Related Info — http://pet.ucla.edu